CLINICAL TRIAL: NCT03643601
Title: A Non-interventional, Epidemiological, Registry-based Evaluation of Anaemia in Swedish Patients With Chronic Kidney Disease (ASK)
Brief Title: A Non-interventional, Epidemiological, Registry-based Evaluation of Anaemia in Swedish Patients With Chronic Kidney Disease
Acronym: ASK
Status: Completed | Type: Observational
Sponsor: Astellas Pharma a/s (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 1517-MA-3139-SN
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Chronic Kidney Disease Associated Anemia
Keywords: erythropoiesis stimulating agent; chronic kidney disease associated anemia; ASP1517

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Dialysis (ND) Patients: For the ND patients, data are captured on each clinic visit during the course of the year (2-4 times per year), the last available record for 2015 will be used.
  Interventions: Other: Non-Interventional
- Dialysis (DD) Patients: For the DD patients, data are input from a randomly selected visit to the hospital in September to October 2015; the evaluation will be based on this record.
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Epidemiological overview of CKD-associated anemia and treatment patterns, rather than to evaluate specific drugs

SUMMARY:
The primary purpose of this study is to describe renal anemia treatment patterns in non-dialysis dependent (ND) and dialysis dependent (DD) populations, with a particular focus on iron use in erythropoiesis stimulating agent (ESA) treated patients.

This study will also provide an epidemiological description of chronic kidney disease (CKD) associated anemia in relation to CKD stage, dialysis modality and underlying morbidity, as well as describe the relationship between inflammation and ESA treatment and describe the associated cardiovascular illness in ESA treated patients.

DETAILED DESCRIPTION:
Data from year 2015 will be used for the prevalence analysis.The prevalent population of CKD patients > 18 years in the Swedish Renal Registry in 2015 both dependent on dialysis (DD) and not on dialysis (ND).

ELIGIBILITY:
Inclusion Criteria:

* For ND-CKD population:

  * all prevalent patients with a CKD with Estimated Glomerular filtration rate (eGFR) < 45ml/min/1.73m2 with a recorded visit pre-dialysis in Swedish Renal Registry (SRR) in 2015
  * Not on dialysis
* For DD-CKD population

  * All prevalent patients taking part in the yearly cross-sectional dialysis investigation in SRR in 2015
  * Dialysis dependent

Exclusion Criteria:

* not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prevalent population of CKD patients > 18 years in the Swedish Renal Registry in 2015 both dependent on dialysis (DD) and not on dialysis (ND); the main analyses will be conducted on patients receiving treatment for renal anaemia.
Sampling Method: Non-Probability Sample
Enrollment: 14415 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
Iron use in erythropoiesis stimulating agent (ESA) treated patients in the prevalent non-dialysis dependent (ND) population | 1 year (data from 2015)
  Route of administration of iron (oral, intravenous (IV), or no iron use) over the source period.
Iron use in ESA treated patients in the prevalent dialysis dependent (DD) population | 1 year (data from 2015)
  Route of administration of iron (oral, intravenous (IV), or no iron use) over the source period.

SECONDARY OUTCOMES:
Proportion of non-dialysis dependent (ND) patients on low, normal, high dose erythropoiesis stimulating agent (ESA) | 1 year (data from 2015)
  The proportion of ND patients on low, normal and high dose ESA will be calculated.
Proportion of dialysis dependent (DD) patients on low, normal, high dose ESA | 1 year (data from 2015)
  The proportion of DD patients on low, normal and high dose ESA will be calculated.
ESA use in ND patients at each CKD stage | 1 year (data from 2015)
  The number of ND patients using/not using ESA at each CKD stage.
ESA use in DD patients | 1 year (data from 2015)
  The number of DD patients using/not using ESA.
Proportion of ND patients treated with ESAs at each chronic kidney disease (CKD) stage with or without oral/IV iron | 1 year (data from 2015)
  Proportion of ND patients treated with ESAs in each CKD stage with or without oral/iv iron.
Proportion of DD patients treated with ESAs at each chronic kidney disease (CKD) stage with or without oral/IV iron | 1 year (data from 2015)
  Proportion of DD patients treated with ESAs in each CKD stage with or without oral/iv iron.
Proportion of ESA treated ND patients within Haemoglobin (Hb) levels within pre-specified target range | 1 year (data from 2015)
  Proportion of ND patients within pre-specified Hb target.
Proportion of ESA treated DD patients within Haemoglobin (Hb) levels within pre-specified target range | 1 year (data from 2015)
  Proportion of DD patients within pre-specified Hb target.
Proportion of ND patients with anemia who are not treated with ESAs | 1 year (data from 2015)
  Proportion of ND patients with anemia not treated with ESAs.
Proportion of DD patients with anemia who are not treated with ESAs | 1 year (data from 2015)
  Proportion of DD patients with anemia not treated with ESAs.
Proportion of ESA treated ND patients with low or medium and high C-reactive protein (CRP) | 1 year (data from 2015)
  Proportion of ND patients with low, medium or high CRP.
Proportion of ESA treated DD patients with low or medium and high CRP | 1 year (data from 2015)
  Proportion of DD patients with low, medium or high CRP.
Proportion of ESA treated ND patients with hyperlipidemia (HDL/LDL) and/or taking lipid lowering preparations | 1 year (data from 2015)
  Proportion of ESA treated ND patients with hyperlipidemia High density lipoprotein / Low density lipoprotein (HDL/LDL) and/or taking lipid lowering drugs.
Proportion of ESA treated DD patients with hyperlipidemia (HDL/LDL) and/or taking lipid lowering preparations | 1 year (data from 2015)
  Proportion of ESA treated DD patients with hyperlipidemia (HDL/LDL) and/or taking lipid lowering drugs.
Proportion of ESA treated ND patients with high blood pressure and/or taking anti-hypertensive medication | 1 year (data from 2015)
  Proportion of ESA treated ND patients with high blood pressure and/or taking anti-hypertensive drugs.
Proportion of ESA treated DD patients with high blood pressure and/or taking anti-hypertensive medication | 1 year (data from 2015)
  Proportion of ESA treated DD patients with high blood pressure and/or taking anti-hypertensive drugs.
Number of ND patients with serious cardiovascular events | 4 years (CV events may be compared from data covering 2012 to 2016)
  The number of ND patients with serious cardiovascular events (i.e., myocardial infarction, heart failure, myocardial ischemia) will be evaluated.
Number of DD patients with serious cardiovascular events | 4 years (CV events may be compared from data covering 2012 to 2016)
  The number of DD patients with serious cardiovascular events (i.e., myocardial infarction, heart failure, myocardial ischemia) will be evaluated.
Number of ND patients with serious thromboembolic events | 1 year (data from 2015)
  The number of ND patients with serious thromboembolic events (i.e. stroke) will be evaluated.
Number of DD patients with serious thromboembolic events | 1 year (data from 2015)
  The number of DD patients with serious thromboembolic events (i.e. stroke) will be evaluated.
All cause mortality: ND | 1 year (data from 2015)
  The number of deaths in the ND population.
All cause mortality: DD | 1 year (data from 2015)
  The number of deaths in the DD population.
Correlation between ESA dose and Hb level in relation to CKD severity (stage 3,4, 5 and DD) | 1 year (data from 2015)
  Scatter plots of ESA dose against hemoglobin level for CKD severity (stage 3, 4, 5 and DD).
Correlation between Haemoglobin (Hb) level and CKD severity: ND | 1 year (data from 2015)
  Box plots of ESA dose against CKD severity (stage 3,4, 5).
Correlation between ESA dose and C-reactive protein (CRP) level: ND | 1 year (data from 2015)
  Scatter plot of ESA dose versus CRP level in ND population.
Correlation between ESA dose and CRP level: DD | 1 year (data from 2015)
  Scatter plot of ESA dose versus CRP level in DD population.
Relationship between ESA dose and occurrence of Cardiovascular (CV) events in ND population | 1 year (data from 2015)
  Box plot of ESA dose in ND patients with or without CV events.
Relationship between Hb level and occurrence of CV events in ND population | 1 year (data from 2015)
  Box plot of Hb level in ND patients with or without CV events.
Relationship between Hb level and occurrence of CV events in DD population | 1 year (data from 2015)
  Box plot of Hb level in DD patients with or without CV events.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Advisor, Study Chair — Astellas Pharma a/s
Locations (1):
- SE46001, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=352